CLINICAL TRIAL: NCT04881123
Title: Randomized, Double-blind, Placebo-controlled, Parallel Groups, Multicenter Pivotal Study Assessing the Efficacy and Safety of 15 mg Twice a Day (BID) of SER150 in Well-controlled Type 2 Diabetic Patients With Diabetic Kidney Disease and Albuminuria in Treatment With an Angiotensin Converting Enzyme Inhibitor or an Angiotensin Receptor Antagonist
Brief Title: SER150 vs Placebo in Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Serodus AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SER150 CL-009
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Kidney Disease
Keywords: SER150; Urine albumin-creatinine ratio; Pivotal study; Type 2 diabetes; Albuminuria
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Albuminuria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SER150 (Experimental): Randomized participants will receive SER150, 15 mg, orally, BID (except on Day 168 where participants will only receive a 15 mg single dose (QD) in the morning)
  Interventions: Drug: SER150
- Placebo (Placebo Comparator): Randomized participants will receive matching placebo, orally, BID (except on Day 168 where participants will only receive a 15 mg single dose (QD) in the morning)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SER150 — Dosage Level(s): 30 mg (1 capsule of 15 mg twice a day - morning and evening) (except on Day 168 where participants will only receive a single dose (QD) in the morning)
  Arms: SER150
Drug: Placebo — Dosage Level(s): Matched placebo (1 capsule twice a day - morning and evening) (except on Day 168 where participants will only receive a single dose (QD) in the morning)
  Arms: Placebo

SUMMARY:
This study is to assess the efficacy and safety of SER150 administered for 24 weeks as a 15 mg twice a day BID dose (except on Day 168 15 mg QD) in participants with type 2 diabetes (T2D) and albuminuria in treatment with either an angiotensin converting enzyme inhibitor (ACEi) or an angiotensin receptor antagonist (ARB).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel groups, multicenter pivotal study assessing the efficacy and safety of 15 mg BID (except on Day 168 15 mg QD) of SER150 in well-controlled adult T2D participants with stable concomitant medications, diabetic kidney disease (DKD) and albuminuria in treatment with an ACEi or an ARB.

The randomized treatment period will be 24 weeks followed by a 4-weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participant has had stable T2D for 3 months prior to screening
* Participant has albuminuria defined by urine UACR ≥ 200 mg/g creatinine as a mean of three independent samples of first urine void of the day
* Participant is receiving stable antidiabetic treatment. Antidiabetic treatment includes all drugs given for the treatment of T2D
* Participant is in treatment with ACEi or ARB, with eGFRcrea lower than 75 mL/minute /1.73 m^2 and above 15 mL/minute/1.73 m^2 (CKD-EPI formula) and will not, in the opinion of the investigator, become a candidate for renal dialysis whilst on the study
* Participant is determined to be overtly healthy as determined by Investigator review of their medical history, physical examination, laboratory tests, and cardiac monitoring. It is anticipated that, whilst some of the participant's results may be different to that of a completely healthy individual, the Investigator will review the participant's individual results to ensure they are as healthy as can be expected give the participant's current health status
* Participant has ASA physical status, health class 2, 3 or 4
* Participant has blood pressure ≤ 160 mmHg systolic, and ≤ 100 mmHg diastolic
* Participant has normal electrocardiogram
* Participant has glycosylated hemoglobin (HbA1c) ≤ 10%
* Participant has prothrombin within normal values
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Acute myocardial infarction within the last 3 months
* Stroke within the last 3 months
* Any major surgery in the last 3 months that in the opinion of the Investigator poses an increased bleeding risk.
* ACR ≤ 200 mg/g creatinine
* Urinary bladder infections within the last 3 months (all other urinary tract infections and vulvovaginitis are excluded)
* Recent history (within the last 6 months) or ongoing liver disease, including viral infections
* Participants with HIV
* Participants with known specific renal diseases different from DKD
* Any bleeding disorder or acute blood coagulation defect
* A history of gastric ulcers or any other organic lesion susceptible to bleeding
* Participant has had a confirmed COVID-19 infection by appropriate laboratory test (PCR or Rapid Antigen Test) within the last 4 weeks prior to screening or on admission
* Participant who had severe course of COVID-19
* Any other condition or clinically relevant abnormal findings in physical examination, laboratory results or ECG during screening period that, in the opinion of the Investigator, may compromise the safety of the participant in the study, reduce the participant's ability to participate in the study, or interfere with evaluation of the study drug
* Change in antidiabetic treatment during last 3 months
* Chronic treatment with nonsteroidal anti-inflammatory drugs or other anti-inflammatory compounds during the last month
* Treatment with anticoagulant drugs
* Participation in another clinical trial of an investigational small molecule, antibody (or medical advice) within 30 days (or 5 half-lives of the drug, whichever is longer [if known]) prior to the start of IP administration on Day 2 (or within 6 months prior to the start of IP administration on Day 1 if the investigational drug was a biologic).
* Alanine aminotransferase or aspartate aminotransferase values exceeding 5 x upper limit of normal (ULN)
* Alkaline phosphatase and/or total bilirubin values exceeding 1.5 x ULN
* HbA1c > 10%
* eGFRcrea ≥75 mL/minute/1.73 m^2 and ≤ 15 mL/minute/1.73 m^2
* Allergy to the active substance or any of the excipients of the drug product
* Pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
A change of urine albumin-to-creatinine ratio (UACR) of > 30% from Baseline to Day 168 | Baseline to Day 168
  The efficacy of 15 mg BID of SER150 with placebo will be compared in well controlled type 2 diabetic participants with DKD, and albuminuria in treatment with an ACEi or an ARB.

SECONDARY OUTCOMES:
Change of UACR from Baseline to Day 168 | Baseline to Day 168
  Efficacy of 15 mg BID of SER150 will be determined in well-controlled type 2 diabetic participants with DKD, and albuminuria in treatment with an ACEi or an ARB.
Time to change of eGFRcrea and eGFRcys ≥ 0.50 mL/min/1.73 m^2 | Baseline to Day 168
  Efficacy of 15 mg BID of SER150 will be determined in well-controlled type 2 diabetic participants with DKD, and albuminuria in treatment with an ACEi or an ARB. eGFRcrea is defined as estimated glomerular filtration rate using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation and eGFRcys is defined as estimated glomerular filtration rate using the CKD-EPI cystatin C equation.
Number of participants with a change in eGFRcrea and eGFRcys | Baseline to Day 168
  Efficacy of 15 mg BID of SER150 will be determined in well-controlled type 2 diabetic participants with DKD, and albuminuria in treatment with an ACEi or an ARB.
Number of participants with a change in eGFRcr-cys | Baseline to Day 168
  Efficacy of 15 mg BID of SER150 will be determined in well-controlled type 2 diabetic participants with DKD, and albuminuria in treatment with an ACEi or an ARB. eGFRcr-cys is defined as estimated glomerular filtration rate using CKD-EPI creatinine-cystatin C equation.
Number of participants with end stage renal disease, any serious cardiovascular events (stroke-acute myocardial infarction-cardiovascular death) and all-cause mortality | Screening (up to 21 days before Day 1). Day 1 and from Day 7 until the Follow-up (Day 196)
  Efficacy of 15 mg BID of SER150 will be determined in well-controlled type 2 diabetic participants with DKD, and albuminuria in treatment with an ACEi or an ARB.
Number of participants with adverse events (AEs) | Screening (up to 21 days before Day 1). Day 1 and from Day 7 until the Follow-up (Day 196)
  Safety/tolerability of 15 mg BID of SER150 will be determined in well-controlled type 2 diabetic participants with DKD, and albuminuria in treatment with an ACEi or an ARB.
PK trough SER150 concentrations (pre-dose) | D7, D28, D56, D84, D112, D140 and D168
  Efficacy, Safety/tolerability of 15 mg BID of SER150 will be determined in well-controlled type 2 diabetic participants with DKD, and albuminuria in treatment with an ACEi or an ARB.

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (8):
  - Liverpool Hospital, Liverpool, New South Wales
  - The AIM Centre (Hunter Diabetes Centre), Merewether, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Southern Adelaide Diabetes and Endocrine Services, Adelaide, South Australia
  - SA Endocrine Research, Keswick, South Australia
  - St Vincent's Hospital, Fitzroy, Victoria
  - Sunshine Hospital, Saint Albans, Victoria
- New Zealand (4):
  - Pacific Clinical Research Clinic Rotorua, Rotorua, Bay of Plenty
  - PCRN Silverdale Medical Centre, Silverdale, Hibiscus Coast
  - Lakeland Clinical Trials Waikato, Hamilton, Waikato Region
  - New Zealand Clinical Research (NZCR), Christchurch

IPD SHARING:
Plan to Share IPD: No